CLINICAL TRIAL: NCT02297867
Title: Adipose-Derived Stem Cells (ADSCs) Injections for Liver Cirrhosis
Brief Title: Clinical Trial Study About Human Adipose-Derived Stem Cells in the Liver Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gwo Xi Stem Cell Applied Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sabrina Huang, China Medical University Beigang Hospital, Gwo Xi Stem Cell Applied Technology Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28113265
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2017-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADSCs (Experimental): One milliliter of cell suspension will be injected intrahepatically under sonographic guidance using a gauge-18 needle.
  Interventions: Drug: ADSCs

INTERVENTIONS:
Drug: ADSCs — autologous ADSCs
  Other Names: hADSCs

SUMMARY:
The aim of the investigators study was to investigate the safety and efficacy of autologous ADSCs for the clinical treatment of liver cirrhosis.

DETAILED DESCRIPTION:
One milliliter of cell suspension will be injected intrahepatically under sonographic guidance using a gauge-18 needle.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis investigators with age 20 to 80 years (both inclusive).
2. Investigators without Mandatory Communicable Disease (HBV, HCV, HIV, syphilis)
3. Investigators without rare disorder
4. Coagulation normalities
5. Investigators without autoimmune disorder
6. Investigators without Acquired Immune Deficiency Syndrome
7. Investigators without cancer
8. Investigators BMI > 15

Exclusion Criteria:

1. Pregnant women
2. Investigators with acute stroke in one month and unconsciousness
3. Investigators with acute myocardial infarction or acute heart failure
4. Investigators with serious liver dysfunction and coagulation dysfunction and ascites mild higher
5. Investigators with acute respiratory failure or pneumonia
6. Kidney Failure: BUN > 50
7. Anemia: Hematocrit < 25
8. Investigators diagnosed with liver cancer or liver metastatic carcinoma
9. Investigators with liver abscess
10. Investigators with acute Hepatitis
11. Investigators with acute infective
12. Liver cirrhosis patients with HBV or HCV
13. Investigators diagnosed with carcinoma and receiving treatment
14. Investigators with Schizophrenia or melancholia
15. Investigators received serious surgical operations in 3 months
16. Investigators unable to control hypertension (SBP > 180 mmHg, DBP > 110 mmHg) or diabetes (AC sugar > 200 mg/dl)
17. Others can't fit into the trial evaluate by investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
MELD | 1-6 month
  MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival. It is calculated according to the following formula:MELD = 3.78[Ln serum bilirubin (mg/dL)] + 11.2[Ln INR] + 9.57[Ln serum creatinine (mg/dL)] + 6.43.

CONTACTS AND LOCATIONS:
Overall Officials: CMU B Hospital, Study Director — China Medical University Beigang Hospital
Locations (2):
- Taiwan (2):
  - China Medical University Beigang Hospital, Taichung, Beigang
  - Gwo Xi Stem Cell Applied Technology Co., Ltd., Hsinchu

IPD SHARING:
Plan to Share IPD: Yes
CRO

REFERENCES:
- [Background] Harn HJ, Lin SZ, Hung SH, Subeq YM, Li YS, Syu WS, Ding DC, Lee RP, Hsieh DK, Lin PC, Chiou TW. Adipose-derived stem cells can abrogate chemical-induced liver fibrosis and facilitate recovery of liver function. Cell Transplant. 2012;21(12):2753-64. doi: 10.3727/096368912X652959. Epub 2012 Jul 5. PMID 22776464